CLINICAL TRIAL: NCT02035332
Title: A Two-Phase Clinical Study of the Minerva AURORA Ablation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minerva Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP0001
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-09

CONDITIONS: Menorrhagia Due to Benign Causes
Keywords: Excessive Uterine Bleeding; Menorrhagia; Endometrial Ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aurora Treatment Arm (Experimental): Endometrial Ablation
  Interventions: Device: Aurora Endometrial Ablation System

INTERVENTIONS:
Device: Aurora Endometrial Ablation System — Ablation of the endometrial lining of the uterus using the Aurora System

SUMMARY:
The primary objective of this study is to evaluate the use of the Aurora Ablation System in reducing menstrual blood loss at 12 months post-treatment. The occurrence of adverse events will be assessed along with an assessment of the reduction of uterine bleeding as measured by a pictorial blood loss assessment chart (PBLAC) or menstrual diary.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory menorrhagia with no definable organic cause (abnormal uterine bleeding)
2. Female subject from age 35 to 50 years
3. Uterine sound measurement of 6.0cm to 10.0cm (external os to internal fundus)
4. A minimum PBLAC score of >150 for 3 months prior to study enrollment; OR, A minimum PBLAC score >150 for one month for women who either

   1. had at least 3 prior months documented failed medical therapy; or
   2. had a contraindication to medical therapy; or
   3. refused medical therapy
5. Premenopausal at enrollment as determined by FSH measurement ≤ 40 IU/ml
6. Not pregnant and no desire to conceive at any time
7. Patient agrees not to use hormonal contraception or any other medical intervention for bleeding during the study
8. Able to provide written informed consent using a form that has been approved by the reviewing IRB/EC
9. Subject agrees to follow-up exams and data collection, including ability to accurately use menstrual diaries
10. Subject who is literate or demonstrates an understanding on how to use menstrual diaries

Exclusion Criteria:

1. Pregnancy or subject with a desire to conceive
2. Complex endometrial hyperplasia as confirmed by histology
3. Presence of active endometritis
4. Active pelvic inflammatory disease
5. Active sexually transmitted disease (STD)
6. Presence of bacteremia, sepsis, or other active systemic infection
7. Active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of the procedure
8. Known/suspected gynecological malignancy within the past 5 years
9. Known clotting defects or bleeding disorders
10. Untreated/unevaluated cervical dysplasia
11. Known/suspected abdominal/pelvic cancer
12. Prior uterine surgery (except low segment cesarean section) that interrupts the integrity of the uterine wall (e.g., transmural myomectomy or classical cesarean section)
13. Previous endometrial ablation procedure
14. Currently on medications that could thin the myometrial muscle, such as long-term steroid use
15. Currently on anticoagulants
16. Abnormal or obstructed cavity as confirmed by hysteroscopy or SIS, specifically:

    1. Septate or bicornuate uterus or other congenital malformation of the uterine cavity
    2. Pedunculated or submucosal myomas distorting the uterine cavity
    3. Polyps likely to be the cause of the subject's menorrhagia
    4. Intramural or subserosal myomas that distort the uterine cavity
17. Presence of an intrauterine device (IUD)
18. Subject currently on hormonal birth control therapy or unwilling to use a non-hormonal birth control post-ablation.
19. Any general health condition which, in the opinion of the Investigator, could represent an increased risk for the subject
20. Any subject who is participating in any other research of an investigational drug or device that has not yet completed the primary endpoint evaluation.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Hungary (3):
  - Szt Imre Hospital, Budapest, Budapest
  - University of Szeged, Szeged, Csongrád megye
  - Kenézy Hospital, Debrecen, Hajdú-Bihar

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the clinical trial at 3 investigational sites in Hungary from May 2011 until October 2011.
Pre-assignment Details: 23 subjects enrolled: 2 subjects excluded based on pre-procedure hysteroscopy findings and did not receive treatment, in 1 subject treatment was attempted but procedure was aborted due to the width of the uterus, the remaining 20 subjects completed study treatment. The protocol ITT population included all subjects in whom treatment was attempted.
Period: Overall Study
Arm/Group | Aurora Treatment Arm
Started | 21 (Treatment Attempted)
Treated | 20 (Treatment Completed)
Completed | 20 (Completed 12 Month Follow-up)
Not Completed | 1
Not completed — Procedure Aborted due to Uterine Width | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Subjects
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 23
PBLAC Score (assessment of menstrual blood loss) [Mean (Standard Deviation); unit: units on a scale] — Pictorial Blood Loss Assessment Chart (PBLAC) is a tool used to assess menstrual blood loss. The PBLAC score takes into account the number of menstrual pads and tampons used as well as amount of saturation. A score of 0 represents no bleeding. Although the PBLAC score does not yield an exact measure of blood loss, it has been found to correlate well with menstrual blood volume. A score greater than 100 is correlated with a blood loss of at least 80 mL.
  units on a scale | 419.2 (152.2)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Menstrual Blood Loss to Normal Levels at 12-months
Description: Number of subjects in whom menstrual blood loss was reduced to normal or below normal levels at 12 months, as measured by a pictorial blood loss assessment chart (PBLAC) score of <=75. A score of 0 represents no bleeding.
Time Frame: 12 Months
Population: Protocol Intent-to-treat population (all subjects in whom the experimental device was attempted to be placed.)
Measure: Number; unit: participants
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 21
participants | 20

2. Secondary Outcome: Procedure Time
Description: Procedure time defined as time from insertion of the Disposable Handpiece to the time of removal.
Time Frame: Day of procedure
Population: Subjects completing treatment
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 20
Minutes | 5.2 (2.1)

3. Post Hoc Outcome: Subjects With Amenorrhea at 12 Months
Description: Amenorrhea at 12 Months- Number of Subjects experiencing no menstrual bleeding
Time Frame: 12 Months
Population: Protocol Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 21
participants | 11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aurora Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aurora Treatment Arm (N=21)
Surgery for Heart Valve Replacement (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aurora Treatment Arm (N=21)
Anesthesia Related (Surgical and medical procedures) | 6 (6)
Bleeding (Reproductive system and breast disorders) | 6 (6)
Pelvic Cramping (non-specific) (Reproductive system and breast disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 1 (1)
Back pain-occasional in middle-back (Musculoskeletal and connective tissue disorders) | 1 (1)
pregnancy- empty sac (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Weakness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No